CLINICAL TRIAL: NCT04678193
Title: COVID-19 Risk Assessment Hospitalization Outcomes Epidemiology Efficacy
Brief Title: COVID-19 Risk Assessment for Hospitalization Outcomes and Epidemiology Efficacy
Acronym: COROMEC
Status: Recruiting | Type: Observational
Sponsor: Aventyn, Inc. (Industry)
Collaborators: Intel Corporation (Industry); Abrazo Health Network (Unknown); Karolinska Institutet (Other); ASU College of Health Solutions (Unknown)
Responsible Party: Sponsor
Other Study IDs: CORAVT 001
Record Dates: First submitted 2020-11-06; First posted 2020-12-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19 PCR positive test and negative or high risk asymptomatic: Patient population COVID-19 infection risk assessment real time epidemiology with 27000 subjects
- COVID19 PCR positive test Stage 1 infection: Patient population of PCR positive COVID-19 Stage 1 infection in registry targeted for ECL-19 treatment for reduced hospitalization with 2700 subjects (10% ECL-19 and 20% Placebo)
  Interventions: Drug: Coromec Registry with ECL-19

INTERVENTIONS:
Drug: Coromec Registry with ECL-19 — Glycocheck to assess Microvascular Score will be used on all patients. An algorithm-based identification of symptoms and objective evidence using care coordination and remote sensor driven technology
  Other Names: Glycocheck
  Groups: COVID19 PCR positive test Stage 1 infection

SUMMARY:
Researchers are creating real-time epidemiology registry to evaluate the efficacy of COVID-19 subject risk assessment scores based on recording of symptoms, biomarkers, chronic illness and mental health assessments with digital technology using wearables and mobile app tools. Researchers aim to study in Phase 1, epidemiological variations in COVID-19 presentation in both PCR positive and negative subjects in the registry. Assessment of variables, predictive modeling of variables that impact severity of COVID-19 positive and negative subjects and assessment of predictors for post COVID-19 complications. In Phase 2, 2700 subjects with COVID-19 positive test will be studied in the intervention group comparing ECL-19 vs placebo with primary end point of hospital admission assessment. Treatment strategy for PCR positive COVID-19 subjects in the registry who are in Stage I of the disease process with ECL-19 drug compared to placebo in reducing hospital admissions

DETAILED DESCRIPTION:
Investigators aim is to create a real time COVID-19 Coromec epidemiology registry to assess the feasibility of monitoring subject infection progress using Vitalbeat digital therapeutics monitoring platform for remote patient monitoring and integrated chronic disease management with mobile app, AI-bot, IoT wearables and cloud computing algorithms developed by health technology company Aventyn, Inc., in collaboration with Intel Corp., clinicians and scientists from Baylor Heart, Abrazo Health, Karolinska Institute, Dignity Health. Coromec registry is a real time epidemiology solution deploying Vitalbeat for pandemic public health stakeholders to enable immediate reporting, assess subject risk prediction for COVID-19 avoiding hospitalization.

The digital health technology aims to assess predictors of risk and predictors of preventing COVID-19, assess what preventive strategies are being used and the efficacy of treatment strategies for avoiding hospitalization. The platform launched globally and is available on the public internet at www.coromec.org

Users can self-report symptoms, mental health assessment, chronic illness status and vital sign measures on a daily basis for risk assessment and preventive treatment with a variety of digital tools by downloading Coromec mobile app, access interactive chatbots and the Coromec real time epidemiology website Researchers aim to study ECL-19 as a drug treatment in stabilizing the endothelium as the first line of approach in COVID 19 positive subjects that may quickly restore their glycocalyx and endothelium thus avoiding hospitalizations and progression of disease with ECL-19

A validated approach would enable vulnerable subjects and communities access to pandemic care. Registry data can assist public health scientists in further studies and enable global registries in future pandemic emergencies to help better understand use of digital tools, intelligent algorithms and predict risk outcomes with targeted novel treatment strategies

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 PCR positive
* COVID-19 PCR negative
* COVID-19 PCR pending
* COVID-19 high risk score

Exclusion Criteria:

* Subjects unwilling to participate in the study before, during or after consent
* Patients considered unreliable by the investigator concerning the requirements for follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unselected patient population of COVID 19 positive infection
Sampling Method: Non-Probability Sample
Enrollment: 27000 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Predictors of post COVID-19 complications and predictors of hospitalization | 1 Day
  Measure COVID-19 infection risk score based on PCR Positive Test
Health symptom score | 1 Day
  Measure COVID-19 infection risk score based on health symptoms
Vital signs SpO2 score | 1 Day
  Measure COVID-19 infection high risk score based on vital signs SpO2 <94%
Vital signs BMI score of 40 kg/m2 | 1 Day
  Measure COVID-19 infection high risk score based on Height 0.15 meters and Weight of 122 Kgs
Chronic Illness score | 1 Day
  Measure COVID-19 infection high risk score based on chronic illness response; Yes on uncontrolled Asthma, COPD, Hypertension, T2DM
Mental health assessment high score >11 on PHQ9 Depression score | 1 Day
  Measure COVID-19 infection risk score based on mental health assessment for Depression
Mental health assessment high score >11 on GAD 7 Anxiety score | 1 Day
  Measure COVID-19 infection risk score based on mental health assessment for Anxiety
Evaluate a treatment strategy with ECL-19 | 1 Day
  Measure hospital admissions in PCR positive COVID 19 subjects within 48 hours who are in Stage I of the disease process

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Vink, PhD, Principal Investigator — Maastricht University; Michael Castro, MD, Principal Investigator — Abrazo Health Network; Kris Vijay, MD, Study Chair — Abrazo Health Network
Locations (3):
- Multiple Locations, Phoenix, Arizona, United States
- Multiple Locations, Bangalore, India
- Multiple Locations, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rovas A, Lukasz AH, Vink H, Urban M, Sackarnd J, Pavenstadt H, Kumpers P. Bedside analysis of the sublingual microvascular glycocalyx in the emergency room and intensive care unit - the GlycoNurse study. Scand J Trauma Resusc Emerg Med. 2018 Feb 14;26(1):16. doi: 10.1186/s13049-018-0483-4. PMID 29444696
- [Background] Weissgerber TL, Garcia-Valencia O, Milic NM, Codsi E, Cubro H, Nath MC, White WM, Nath KA, Garovic VD. Early Onset Preeclampsia Is Associated With Glycocalyx Degradation and Reduced Microvascular Perfusion. J Am Heart Assoc. 2019 Feb 19;8(4):e010647. doi: 10.1161/JAHA.118.010647. PMID 30764695
- [Background] Rovas A, Seidel LM, Vink H, Pohlkotter T, Pavenstadt H, Ertmer C, Hessler M, Kumpers P. Association of sublingual microcirculation parameters and endothelial glycocalyx dimensions in resuscitated sepsis. Crit Care. 2019 Jul 24;23(1):260. doi: 10.1186/s13054-019-2542-2. PMID 31340868